CLINICAL TRIAL: NCT02695420
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Omecamtiv Mecarbil in Japanese Subjects With Heart Failure With Reduced Ejection Fraction
Brief Title: Safety, PK, and Efficacy of Omecamtiv Mecarbil in Japanese Subjects With Heart Failure With Reduced Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120227
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo BID (Placebo Comparator): Participants will receive placebo BID.
  Interventions: Drug: 25 mg Omecamtiv Mecarbil
- 25 mg Omecamtiv Mecarbil BID (Experimental): Participants will receive 25 mg omecamtiv mecarbil BID.
  Interventions: Drug: Placebo
- 37.5 mg Omecamtiv Mecarbil BID Target Dose (Experimental): Participants will receive omecamtiv mecarbil 25 mg BID up to Week 4 or Week 8 and 25 mg or 37.5 mg BID after Week 4 or Week 8, based on Week 2 PK.
  Interventions: Drug: 25 mg Omecamtiv Mecarbil; Drug: 37.5 mg Omecamtiv Mecarbil
- 50 mg Omecamtiv Mecarbil BID Target Dose (Experimental): Participants will receive Omecamtiv Mecarbil 25 mg BID up to Week 4 or Week 8 and 25 mg or 50 mg BID after Week 4 or Week 8, based on Week 2 PK.
  Interventions: Drug: 25 mg Omecamtiv Mecarbil; Drug: 50 mg Omecamtiv Mecarbil

INTERVENTIONS:
Drug: 25 mg Omecamtiv Mecarbil — oral tablet
  Arms: 37.5 mg Omecamtiv Mecarbil BID Target Dose; 50 mg Omecamtiv Mecarbil BID Target Dose; Placebo BID
Drug: Placebo — oral tablet
  Arms: 25 mg Omecamtiv Mecarbil BID
Drug: 37.5 mg Omecamtiv Mecarbil — oral tablet
  Arms: 37.5 mg Omecamtiv Mecarbil BID Target Dose
Drug: 50 mg Omecamtiv Mecarbil — oral tablet
  Arms: 50 mg Omecamtiv Mecarbil BID Target Dose

SUMMARY:
* To evaluate pharmacokinetics (PK) of omecamtiv mecarbil in Japanese subjects with heart failure (HF) with reduced ejection fraction
* To evaluate the safety and tolerability of oral omecamtiv mecarbil

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female ≥ 20 years and ≤ 85 years of age
* History of chronic stable heart failure (HF) with reduced ejection fraction, defined as requiring treatment for HF for a minimum of 4 weeks prior to screening
* Treated for HF with optimal pharmacological therapy
* Left ventricular ejection fraction ≤ 40% at screening

Exclusion Criteria:

* Severe uncorrected valvular heart disease
* Hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, or clinically significant congenital heart disease
* Acute myocardial infarction, unstable angina, or persistent angina at rest within 30 days prior to randomization
* Systolic blood pressure (BP) > 160 mmHg or < 90 mmHg, or diastolic BP > 90 mmHg, or heart rate (HR) > 110 beats per minute (bpm) or HR < 50 bpm
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2
* Total bilirubin (TBL) ≥ 2x upper limit of normal (ULN), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3x ULN Other Exclusion Criteria may apply.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (27):
- Japan (27):
  - Research Site, Kasugai-shi, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Asahi-shi, Chiba
  - Research Site, Chiba, Chiba
  - Research Site, Imabari, Ehime
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Hakodate-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki-shi, Hyōgo
  - Research Site, Kawanishi-shi, Hyōgo
  - Research Site, Takarazuka-shi, Hyōgo
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Nankoku-shi, Kochi
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Kishiwada-shi, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Saitama-shi, Saitama
  - Research Site, Wako-shi, Saitama
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Meguro-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 31 research centers in Japan from 14 April 2016 to 16 December 2016.
Pre-assignment Details: Participants were randomized at a ratio of 1:1:1:1 to twice daily (BID) placebo, 25 mg, 25 mg->37.5 mg Target Dose, or 25 mg->50 mg Target Dose, respectively. Randomization was stratified by presence or absence of atrial fibrillation/flutter.
Groups:
- Placebo BID: Placebo for omecamtiv mecarbil BID
- Omecamtiv Mecarbil 25 mg BID: Omecamtiv mecarbil 25 mg BID
- Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose: Omecamtiv mecarbil 25 mg BID up to Week 4 or Week 8 and 25 mg or 37.5 mg BID after Week 4 or Week 8, based on Week 2 PK
- Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose: Omecamtiv Mecarbil 25 mg BID up to Week 4 or Week 8 and 25 mg or 50 mg BID after Week 4 or Week 8, based on Week 2 PK
Period: Overall Study
Arm/Group | Placebo BID | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose
Started | 21 | 21 | 19 | 20
Completed | 21 | 20 | 19 | 20
Not Completed | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose | Total
Number analyzed (Participants) | 21 | 21 | 19 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.5) | 66.9 (10.3) | 63.6 (10.8) | 66.5 (12.2) | 65.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 0 | 1 | 13
  Male | 12 | 18 | 19 | 19 | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 21 | 21 | 19 | 20 | 81
  Other | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 21 | 21 | 19 | 20 | 81
  Other | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation/Flutter at Randomization [Number; unit: participants] — Randomization was stratified by presence or absence of atrial fibrillation/flutter via interactive voice-response system/interactive web-response (IVRS/IWRS) system.
  participants
    Present | 4 | 4 | 3 | 4 | 15
    Absent | 17 | 17 | 16 | 16 | 66

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Concentration Before Morning Dose (Cpredose) Over Time
Time Frame: Before morning dose on Week 2 (Day 15), Week 4 (Day 28), Week 12 (Day 84), Week 16 (Day 112)
Population: PK Analysis Set: all randomized participants who received at least one dose of omecamtiv mecarbil and had at least one evaluable omecamtiv mecarbil PK concentration at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose
Number analyzed (Participants) | 20 | 18 | 20
ng/mL
  Week 2 | 239 (106) | 179 (77.1) | 208 (61.6)
  Week 4: number analyzed (Participants) | 17 | 17 | 20
  Week 4 | 222 (63.5) | 196 (44) | 209 (61.9)
  Week 12: number analyzed (Participants) | 19 | 17 | 19
  Week 12 | 217 (66.1) | 228 (56.9) | 282 (120)
  Week 16: number analyzed (Participants) | 19 | 17 | 20
  Week 16 | 206 (84.5) | 244 (67.7) | 292 (118)

2. Primary Outcome: PK: Area Under the Curve Until 8 Hours After Morning Dose at Week 8 (AUC0-8)
Time Frame: Week 8 (Day 56) at predose, at 2 hours ±30 minutes; 4 hours ±30 minutes; 6 hours ±30 minutes; 8 hours ±30 minutes after morning dose
Population: PK Analysis Set: all randomized participants who received at least one dose of omecamtiv mecarbil and had at least one evaluable omecamtiv mecarbil PK concentration.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose
Number analyzed (Participants) | 9 | 8 | 1
hr*ng/mL | 1850 (563) | 1850 (383) | 2360 (465)

3. Secondary Outcome: Change From Baseline at Week 16 in Systolic Ejection Time (SET)
Description: LS mean was from the repeated measures model, which included treatment group, stratification factor (from IVRS), scheduled visit, baseline value, and the interaction of treatment group with scheduled visit as covariates.
Time Frame: Baseline, Week 16 (Day 112)
Population: All participants who received at least one dose of study drug with observed data. The 4 active treatment arms include only those participants who had a minimum investigational product exposure period of 25 days.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Placebo BID | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose
Number analyzed (Participants) | 20 | 19 | 17 | 17
msec | -1.7 (4.7) | 20.5 (4.9) | 27.6 (5.4) | 23.8 (5.2)
Statistical Analysis 1: Comparison: Placebo BID vs Omecamtiv Mecarbil 25 mg BID; Test type: Superiority; p = 0.0008, Repeated Measures Model; Treatment Difference = 22.1, 95% CI 2-sided [9.6 to 34.7], Standard Error of Mean 6.3
Statistical Analysis 2: Comparison: Placebo BID vs Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose; Test type: Superiority; p < 0.0001, Repeated measures model; Treatment Difference = 29.3, 95% CI 2-sided [16.3 to 42.3], Standard Error of Mean 6.5
Statistical Analysis 3: Comparison: Placebo BID vs Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose; Test type: Superiority; p = 0.0002, Repeated measures model; Treatment Difference = 25.5, 95% CI 2-sided [12.6 to 38.4], Standard Error of Mean 6.5

4. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence. Serious AEs are defined as AEs that meets at least 1 of the following serious criteria: fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, other medically important serious event. AEs are graded as: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death. TEAEs are defined as events occurring after the first dose of study drug.
Time Frame: From first dose of study drug up to Week 20 (Day 140 + 3 days)
Population: Safety Analysis Set: all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose
Number analyzed (Participants) | 21 | 21 | 19 | 20
Participants
  All TEAEs | 14 | 10 | 10 | 12
  Grade >= 2 TEAEs | 10 | 6 | 6 | 7
  Grade >= 3 TEAEs | 3 | 4 | 1 | 2
  Grade >= 4 TEAEs | 0 | 1 | 0 | 0
  Serious AEs | 3 | 4 | 1 | 3
  TEAEs Leading to Withdrawal of Study Drug | 0 | 2 | 1 | 0
  Fata Adverse Events | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 20 (Day 140 + 3 days)
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo BID | Omecamtiv Mecarbil 25 mg BID | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/21 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/21 | 4/21 | 1/19 | 3/20
Other Adverse Events (participants affected / at risk) | 10/21 | 8/21 | 10/19 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID (N=21) | Omecamtiv Mecarbil 25 mg BID (N=21) | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose (N=19) | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose (N=20)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Vascular stent restenosis (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID (N=21) | Omecamtiv Mecarbil 25 mg BID (N=21) | Omecamtiv Mecarbil 25 mg to 37.5 mg BID Target Dose (N=19) | Omecamtiv Mecarbil 25 mg to 50 mg BID Target Dose (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 2 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 1 | 4 | 4
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Protein urine (Investigations) | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT02695420/Prot_002.pdf
  • Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02695420/SAP_001.pdf